CLINICAL TRIAL: NCT06760143
Title: Antibiotic Prophylaxis in Lung-Transplant Recipients: a Retrospective Cohort Study
Brief Title: Antibiotic Prophylaxis in Lung-Transplant Recipients
Acronym: PRO-LUNG
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PRO-LUNG
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-10

CONDITIONS: Lung-transplant Recipients; Antibiotic Prophylaxis
Keywords: Lung-Transplant Recipients; piperacillin/tazobactam; levofloxacin; bacterial infections; Multi Drug Resistant Organisms
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients underwent Lung Transplant (LT) and received peri-operative antibiotic prophylaxis: All adult (≥ 18 years) patients who underwent Lung Transplant (LT) and received peri-operative antibiotic prophylaxis.

SUMMARY:
Retrospective, monocentric observational pharmacological cohort study including all adult patients who underwent lung transplantation at IRCCS Azienda Ospedaliero-Universitaria di Bologna from 1st January 2002 to 31st August 2023.

DETAILED DESCRIPTION:
Bacterial infections are clinically relevant complications in lung transplant recipients (LTRs) causing chronic lung allograft dysfunction and high rates of mortality, especially within the first year after transplant. Microorganisms responsible for infection can derive from the donor lung or pre-existing recipient flora. Indeed, even though native lungs are removed, colonization of the grafts from recipients colonizing strains often rapidly occurs.

Furthermore, grafts and preservation fluids are frequently infected or colonized with bacteria with a high transmissibility rate to LTRs.

The interpretation of bacterial growth from grafts and preservation fluids can be complex. While some experts recommend against using lungs that show growth of gram-negative bacteria, others permit their use if accompanied by targeted antibiotic therapy, citing retrospective studies that suggest similar overall survival rates for recipients of infected versus uninfected lungs. To prevent donor-derived infections, routine antibiotic prophylaxis is used. International guidelines recommendations are generic and predominantly based on cardiac procedures and no formal recommendations to guide antimicrobial selection in lung transplant (LT) surgery are currently available. Therefore, antibiotic regimens for perioperative prophylaxis are based on clinical judgment and knowledge of the local epidemiology, inducing heterogeneity in clinical practice between centers. In our Center, for the last 20 years, piperacillin/tazobactam plus levofloxacin has been the backbone of the antibiotic prophylaxis regimen for LTRs, according to internal guidelines.

This retrospective observational study aims to investigate the efficacy of piperacillin/tazobactam plus levofloxacin compared to piperacillin/tazobactam alone as antibiotic prophylactic regimens on preventing early bacterial infections and donor derived infection after LT and their possible impact on subsequent colonization by MDR organisms (MDRO). With the study, it will be possible to evaluate which of the two analyzed regimens is associated with a better outcome in the LTR cohort in terms of preventing early surgical site infections, covering the susceptibility of isolates from donor cultures, and influencing MDRO colonization. In this way, it will be possible to influence clinical practice in the center, improving the prognosis of patients undergoing LT. Finally, the data obtained from this study will contribute to increase the knowledge on prophylaxis regimens that can be adopted in hospitals with a similar epidemiological scenario.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥ 18 years)
* Patients who underwent LT at IRCCS Azienda Ospedaliero-Universitaria di Bologna from 1st January 2002 to 31st August 2023
* Patients receiving peri-operative antibiotic prophylaxis according to internal guidelines at time of LT
* Signed informed consent

Exclusion Criteria:

* Lack of clinical and/or laboratory data regarding type of early bacterial infection and/or antibiotic prophylaxis received after lung transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult (≥ 18 years) patients who underwent Lung Transplant (LT) and received peri-operative antibiotic prophylaxis during the study period will be screened for inclusion. Patients are enrolled during follow-up visits within 5 months from the start of the study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Diagnosis of early postoperative infections and/or bacterial donor-derived infections | Retrospective recruitment period will span from January 2001 to August 2023, with a 60-day retrospective follow-up post-transplant
  Diagnosis of early postoperative infections and/or donor-derived bacterial infections acquired within 15 days of lung transplantation. This is expressed as a four-group composite endpoint: no infection, early postoperative infections only, donor-derived bacterial infections only, both early postoperative and donor-derived bacterial infections

SECONDARY OUTCOMES:
Rectal, urinary and/or respiratory colonization rates by MDRO | Retrospective recruitment period will span from January 2001 to August 2023, with a 60-day retrospective follow-up post-transplant
  Rectal, urinary and/or respiratory colonization rates by MDRO within 60 days from transplant
Susceptibility or resistance to piperacillin/tazobactam and/or levofloxacin | Retrospective recruitment period will span from January 2001 to August 2023, with a 60-day retrospective follow-up post-transplant
  Susceptibility or resistance to piperacillin/tazobactam and/or levofloxacin defined according to each pathogen's breakpoint on MIC values

CONTACTS AND LOCATIONS:
Overall Officials: Renato Pascale, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- Irccs Aoubo, Bologna, Italy